CLINICAL TRIAL: NCT02592720
Title: Intracoronary Cocktail Injection Improves Outcomes of Fractional Flow Reserve Guided Percutaneous Coronary Intervention in Patients With Acute Coronary Syndrom (ACS)
Brief Title: Cocktail Injection Improves Outcomes of FFR Guided PCI
Acronym: CocktailII
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, sunddong, Principal Investigator, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cocktail II-FFR ACS
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes; Fractional Flow Reserve; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Tirofiban; bivalirudin; Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cocktail plus FFR guided group (Experimental): Intracoronary cocktail injection before fractional flow reserve (FFR) measurement. Percutaneous Coronary Intervention (PCI) strategy is decided by FFR value in patients with acute coronary syndrome (ACS).
  Interventions: Drug: cocktail; Device: FFR
- QCA guided group (Placebo Comparator): Percutaneous Coronary Intervention (PCI) strategy is decided by QCA value in patients with acute coronary syndrome (ACS).
  Interventions: Device: QCA guided group

INTERVENTIONS:
Drug: cocktail — Intracoronary cocktail injection before fractional flow reserve (FFR) measurement. Percutaneous Coronary Intervention (PCI) strategy is decided by FFR value in patients with acute coronary syndrome (ACS).
  Other Names: cocktail (tirofiban, bivalirudin, tenecteplase)
  Arms: Cocktail plus FFR guided group
Device: FFR — Percutaneous Coronary Intervention (PCI) strategy is decided by FFR value in patients with acute coronary syndrome (ACS).
  Other Names: pressure wire (St. Jude Medical, Inc.)
  Arms: Cocktail plus FFR guided group
Device: QCA guided group — Percutaneous Coronary Intervention (PCI) strategy is decided by QCA value in patients with acute coronary syndrome (ACS).
  Arms: QCA guided group

SUMMARY:
This is a randomized, single blind, controlled study of intracoronary cocktail injection before fractional flow reserve (FFR) measurement when guiding percutaneous coronary intervention (PCI) in patients with acute coronary syndrome (ACS).

DETAILED DESCRIPTION:
This is a randomized, single blind, controlled study of intracoronary cocktail injection before fractional flow reserve (FFR) measurement when guiding percutaneous coronary intervention (PCI) in patients with acute coronary syndrome (ACS). Patients with ACS will be randomized into the cocktail plus FFR guided group or the QCA guided group. The primary outcome of the cocktail II study is the composite of death, myocardial infarction, class IV heart failure and target vessel revascularization within 1 year. The secondary outcome of the cocktail II study include left ventricular function, quality of life, stroke or life-threatening bleeding within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* patients with a clinical diagnosis of recent ACS within 5 days

Exclusion Criteria:

* haemodynamic instability
* intolerance to anti-platelet drugs
* ineligible for coronary revascularization
* a treatment plan for non-coronary heart surgery (e.g. valve surgery)
* a history of prior PCI or CABG
* angiographic evidence of severe (e.g. diffuse calcification) or mild (<30% severity) coronary disease
* a life expectancy less than 1 year
* adenosine allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 1 year
  number of participants with death, myocardial infarction or class IV heart failure and target vessel revascularization revascularization

SECONDARY OUTCOMES:
left ventricular function | 1 year
  left ventricular ejection fraction evaluated by ultrasound and MRI
Seattle Angina Questionnaire scores | 1 year
  Seattle Angina Questionnaire scores
Canadian Cardiovascular Society (CCS) Functional Angina classification | 1 year
  Canadian Cardiovascular Society (CCS) Functional Angina classification
6-minute walk distance (6MWD) | 1 year
  6-minute walk distance (6MWD)
stroke | 1 year
  number of participants with stroke

CONTACTS AND LOCATIONS:
Overall Officials: Dongdong Sun, M.D.,Ph.D., Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China